CLINICAL TRIAL: NCT04743076
Title: Standard Medical Treatment Plus Endovascular Treatment Versus Standard Medical Treatment Alone for Stroke Patient With Large Vessel Occlusion In The Posterior Circulation: A Multicenter, Randomized, Clinical Trial
Brief Title: A Randomized Trial Of Endovascular Treatment For Acute Posterior Large Vessel Occlusion
Acronym: BASILAR-2
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawal of funding
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BASILAR-2
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Vertebrobasilar Stroke
Keywords: endovascular treatment; thrombolysis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Standard medical treatment plus endovascular treatment
  Interventions: Procedure: Endovascular treatment; Other: Standard medical treatment
- Control group (Active Comparator): Standard medical treatment alone
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Procedure: Endovascular treatment — Endovascular treatment
  Arms: Intervention group
Other: Standard medical treatment — Standard medical treatment

SUMMARY:
The aim of this trial is to investigate whether endovascular treatment can improve the 90-day functional outcome of acute large vessel occlusion in the posterior circulation.

DETAILED DESCRIPTION:
At least seven randomized controlled trials have consistently shown that endovascular treatment can improve the functional outcome of stroke patients with acute anterior large vessel occlusion. However, these trials did not include patients with large vessel occlusion in the posterior circulation.

The hypothesis of this trial: Compared with standard medical treatment alone, standard medical treatment combined with endovascular treatment can significantly improve the 90-day functional outcome of acute large vessel occlusion in the posterior circulation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: i. 18 ~ 80 years old, pc-ASPECTS score ≥ 6; ii. > 80 years old, pc-ASPECTS score ≥ 8 and mRS = 0 before the onset
2. NIHSS score ≥ 10 before randomization;
3. VA-V4 or basilar artery occlusion proved by CTA/MRA/DSA;
4. Time from stroke onset to randomization within 23.5 hours;
5. Written informed consent is obtained from patients and/or their legal representatives.

Exclusion Criteria:

1. CT or MR evidence of intracranial hemorrhage;
2. Pre-morbidity with a modified Rankin scale score ≥ 3;
3. The patient is in deep coma;
4. Currently in pregnant or lactating or serum beta HCG test is positive on admission;
5. Arterial tortuosity and/or other arterial disease that would prevent the device from reaching the target vessel;
6. Contraindication to radiographic contrast agents, nickel, titanium metals or their alloys;
7. Significant mass effect in the cerebellar hemisphere or hydrocephalus on imaging;
8. Imaging manifestations of diffuse bilateral brainstem ischemia;
9. Multivessel occlusive disease (combined with anterior and posterior circulation occlusion or subtotal occlusion);
10. Cerebral vasculitis, intracranial arteriovenous malformation, aneurysm, or brain tumor with mass effect;
11. Participating in other clinical trials;
12. Any terminal illness with life expectancy less than 6 months;
13. Patients with a preexisting neurological or psychiatric disease that would confound the neurological functional evaluations;
14. Past neurological or psychiatric diseases that hinder the assessment of neurological function;
15. Unlikely to be available for 90-day follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-05-16 (Estimated); Study Completion 2024-05-16 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale score | 90 days
  disability level

SECONDARY OUTCOMES:
Rate of a score of 0~2 on modified Rankin scale | 90 days
  Functional independence
Improvement in NIHSS between baseline and 24 hours | at 24 hours from randomization
  neurological changes
Improvement in NIHSS between baseline and 5~7d | at 5~7 days from randomization
  neurological changes
Improvement in GCS between baseline and 24 hours | at 24 hours from randomization
  neurological changes
Improvement in GCS between baseline and 24 hours | at 5~7 days from randomization
  neurological changes
Asymptomatic intracranial hemorrhage within 48 hours | within 48 hours after endovascular treatment
  evaluate intracranial hemorrhage
Procedural-related complications and severe adverse events | within 90 days
  evaluate complications and any adverse events
Serious non-hemorrhagic adverse events | within 90 days
  evaluate complications and any adverse events
Score of 90-day EQ-5D scale | 90 days
  Functional independence
Mortality within 90 days | 90 days
  evaluate death rate of the two treatment groups
Symptomatic intracranial hemorrhage within 48 hours | within 48 hours after endovascular treatment
  evaluate intracranial hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Qingwu Yang, MD, Principal Investigator — Neurology, Xinqiao Hospital of the Army Medical University; Wenjie Zi, MD, Principal Investigator — Neurology, Xinqiao Hospital of the Army Medical University; Raul G Nogueira, MD, Principal Investigator — Marcus Stroke & Neuroscience Center, Grady Memorial Hospital, Emory University, Atlanta, USA; Jeffrey L Saver, MD, Principal Investigator — Neurology, University of California, Los Angeles, USA
Locations (16):
- China (16):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Banan District People's Hospital, Banan, Chongqing Municipality
  - Xinqiao Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - Wuyi Traditional Chinese Medicine Hospital, Jiangmen, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Maoming Traditional Chinese Medicine Hospital, Maoming, Guangdong
  - Chinese Medical Hospital of Zhongshan, Zhongshan, Guangdong
  - The 924th Hospital of CPLA, Guilin, Guangxi
  - Danzhai People's Hospital, Longquan, Guizhou
  - Nanyang Central Hospital, Nanyang, Henan
  - Wuhan No. 1 Hospital, Wuhan, Hubei
  - The 904th Hospital of CPLA, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
study data without patient information
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Related papers published 3 months later, the IPD will be shared
Access Criteria: yangqwmlys@163.com ziwenjie1981@163.com

REFERENCES:
- [Result] Writing Group for the BASILAR Group; Zi W, Qiu Z, Wu D, Li F, Liu H, Liu W, Huang W, Shi Z, Bai Y, Liu Z, Wang L, Yang S, Pu J, Wen C, Wang S, Zhu Q, Chen W, Yin C, Lin M, Qi L, Zhong Y, Wang Z, Wu W, Chen H, Yao X, Xiong F, Zeng G, Zhou Z, Wu Z, Wan Y, Peng H, Li B, Hu X, Wen H, Zhong W, Wang L, Jin P, Guo F, Han J, Fu X, Ai Z, Tian X, Feng X, Sun B, Huang Z, Li W, Zhou P, Tu M, Sun X, Li H, He W, Qiu T, Yuan Z, Yue C, Yang J, Luo W, Gong Z, Shuai J, Nogueira RG, Yang Q. Assessment of Endovascular Treatment for Acute Basilar Artery Occlusion via a Nationwide Prospective Registry. JAMA Neurol. 2020 May 1;77(5):561-573. doi: 10.1001/jamaneurol.2020.0156. PMID 32080711